CLINICAL TRIAL: NCT01649141
Title: National Child Traumatic Stress Initiative: Community Treatment and Service Centers
Brief Title: Trauma-Focused Cognitive Behavior Therapy for Youth: Effectiveness in a Community Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Delaware Division of Prevention and Behavioral Health Services (Other Government)
Collaborators: University of Medicine and Dentistry of New Jersey (Other); University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SM57145
Record Dates: First submitted 2012-07-19; First posted 2012-07-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: posttraumatic stress disorder; trauma-focused cognitive behavioral therapy; trauma; child abuse
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): Trauma-Focused Cognitive Behavioral Therapy
  Interventions: Behavioral: Trauma-Focused Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Trauma-Focused Cognitive Behavioral Therapy — Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) is a structured, 12-16 session outpatient intervention originally developed to treat Posttraumatic Stress Disorder (PTSD) and related emotional and behavioral difficulties in youth with a history of child sexual abuse. TF-CBT's eight components are delivered in 90-minute weekly sessions split evenly between children and their parents. These components are summarized by the acronym PRACTICE including: psychoeducation and parenting skills (P), relaxation (R), affective expression and regulation (A), cognitive coping (C), trauma narrative development and processing (T), in vivo gradual exposure (I), conjoint parent/child sessions (C) and enhancing safety and future development (E).

SUMMARY:
This effectiveness study is being conducted to determine whether Trauma-Focused Cognitive Therapy (TF-CBT), a treatment model developed in specialty clinics by experts in the treatment of child sexual abuse, can be effectively transported to a state-contracted community mental health agency in the state of Delaware and used effectively by clinicians with little prior TF-CBT experience. The sample is comprised of youths receiving public mental health services and with diverse trauma histories.

DETAILED DESCRIPTION:
This investigation aims to examine the effectiveness of Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) in treating child traumatic stress when implemented in community settings on a state-wide level in Delaware. Youth (ages 7-16 years) with a history of documented trauma (sexual or physical abuse, traumatic loss, domestic or community violence) and symptoms of Posttraumatic Stress Disorder (PTSD) receive approximately 10 sessions of TF-CBT delivered in a state-contracted mental health agency. Children and adolescents are recruited from a public mental health population. PTSD symptoms and internalizing and externalizing behavior problems have been assessed in the first 72 participants at pre-treatment and then at 3-, 6-, 9-, and 12-months after intake; subsequent participants (n=38) are only being assessed for symptoms and problems at pre-treatment and then at 3-, 6-months after intake.

ELIGIBILITY:
Inclusion Criteria:

* child is 7-17 years old
* positive screen for PTSD
* child qualifies for public insurance
* parent willing to co-participate in treatment
* English-speaking (child and parent)

Exclusion Criteria:

* intellectual disability (child)
* untreated psychosis (child)
* untreated substance abuse (child)
* sibling already in study
* unable to participate in year-long follow-up (e.g., moving out of state)

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2006-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change in baseline PTSD Symptoms at 3-,6-,9- and 12-months | Baseline and post-baseline (3-,6-,9-,12-months)
  PTSD symptoms area assessed with the UCLA PTSD Reaction Index for DSM-IV (UPID). The UPID (Pynoos, et al., 1998) includes 48 items that can be administered as a questionnaire or structured interview. The instrument's three sections assess for trauma exposure and symptoms of DSM-IV PTSD in children ages 7-18. The UPID has good convergent validity (i.e., 0.70 in comparison to the K-SADS, epidemiologic version), a sensitivity of 0.93 and specificity of 0.87 in diagnosing PTSD (Steinberg et al., 2004), and test-retest reliability of 0.84 (Steinberg et al., 2004)

SECONDARY OUTCOMES:
Change in baseline behavioral problems at 3-, 6-, 9- and 12-months. | Baseline and post-baseline (3-,6-,9-,12-months)
  Behavioral problems are assessed with the parent version of the Child Behavior Checklist 6-18 (CBCL: Achenbach, & Rescorla, 2001)\.The CBCL is a 113-item parent self-report measure used to assess children's emotional and behavioral problems and social competencies. The CBCL has been used with acceptable levels of reliability (range 0.84-0.98) and content and criterion validity to measure mental health problems of children ages 6-18 years from diverse racial and ethnic backgrounds (Achenbach & Rescorla, 2001).

CONTACTS AND LOCATIONS:
Overall Officials: Charles P Webb, Ph.D., Study Director — Division of Prevention and Behavioral Health Services; Nancy Widdoes, M.A., Principal Investigator — Division of Prevention and Behavioral Health Services
Locations (1):
- Division of Prevention and Behavioral Health Services, Wilmington, Delaware, United States